CLINICAL TRIAL: NCT06456840
Title: Determination of Risk Factors of Shoulder Pathologies in Parkinson Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 24277
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease; Shoulder Pain
MeSH Terms: conditions — Parkinson Disease; Shoulder Pain | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: 40 Parkinson's patients who described pain in at least one shoulder (VAS>3)
  Interventions: Diagnostic Test: ULTRASOUND
- Group 2: 0 Parkinson's patients with undefined pain in both shoulders (VAS: 0)
  Interventions: Diagnostic Test: ULTRASOUND
- Group 3: 40 patients of similar age and gender, without a Parkinson's diagnosis, with any shoulder pain (VAS>3)
  Interventions: Diagnostic Test: ULTRASOUND
- Group 4: 40 patients of similar age and gender, diagnosed without Parkinson's disease and without pain in both shoulders (VAS: 0)
  Interventions: Diagnostic Test: ULTRASOUND

INTERVENTIONS:
Diagnostic Test: ULTRASOUND — Measurements will be made in musculoskeletal system ultrasonography by an international Medicine and Rehabilitation assistant physician using images obtained with the Sonosite M-Turbo device using the ImageJ program. During the measurements, the patient and the patient will be face to face and the device will be placed postero-laterally. Five standard window spacings will be used for the shoulder attachment. These are: anterior transverse, anterior longitudinal, lateral longitudinal, lateral transverse, posterior transverse.

SUMMARY:
Parkinson's disease was first described in history in 1817 by James Parkinson in his monograph "An essay on swinging palsy", and today it is the 2nd most common neurodegenerative disease after Alzheimer's, affecting approximately 6.1 million people. Its main histopathological feature is the decrease in dopaminergic secretion in the basal ganglia and there are three cardinal findings: Bradykinesia, Tremor, Rigidity. Although joint and skeletal deformities are seen in approximately 70% of Parkinson's patients, they are not adequately evaluated and cause significant functional disability and chronic pain, independent of motor symptoms.Musculoskeletal pathologies seen in Parkinson's patients can be classified as: musculoskeletal pain, articular problems, postural problems and bone mineralization defects. The shoulder girdle is a joint with complex and delicate function, consisting of four joints (glenohumeral, sternoclavicular, acromioclavicular and scapulothoracic), supporting muscles and periarticular ligaments, which seriously affects the patient's quality of daily life and function. Although magnetic resonance imaging (MRI) is the best imaging tool in the diagnosis of musculoskeletal system pathologies, it is quite sensitive to artifact-forming motion. Ultrasound (US) imaging is widely used in the evaluation of rotator cuff muscles, biceps muscle and glenohumeral joint pathologies and has many advantages over MRI, such as providing fast, cheap and dynamic imaging. Although many studies have proven that shoulder girdle musculoskeletal pathologies such as bicipital tendinitis, m.supraspinatus tendinosis, subacromial/subdeltoid bursitis, subacromial impingement syndrome, and adhesive capsulitis are seen more frequently in Parkinson's patients by ultrasonographic imaging, these shoulder girdle pathologies seen in Parkinson's patients are more common. The risk factors for pathologies have not been defined. In this study, we aimed to determine the ultrasonographic findings and risk factors of shoulder pathologies in Parkinson's patients and to investigate the effects of shoulder pathologies on quality of daily life, physical activity, falls and balance.

ELIGIBILITY:
Inclusion Criteria:

Group1

* Being diagnosed with Parkinson's according to the Movement Disorders Society diagnostic criteria
* Being over 50 years old
* Being in the Hoehn & Yahr stage I-IV range
* Identification of pain in at least one shoulder (VAS>3)
* Agreeing to participate in the study
* Being literate

Group2

* Being diagnosed with Parkinson's according to the Movement Disorders Society diagnostic criteria
* Being over 50 years old
* Being in the Hoehn & Yahr stage I-IV range
* No pain in both shoulders (VAS: 0)
* Agreeing to participate in the study
* Being literate

Group 3

* Describe pain >3 on the visual pain scale in any shoulder
* Being over 50 years old
* Becoming literate
* Agreeing to participate in the study

Group 4

1. Not defining pain with a score of 0 on the visual pain scale in both shoulders
2. Being over 50 years old
3. Being literate
4. Agreeing to participate in the study

Exclusion Criteria:

* Scoring less than 24 points in the Mini Mental Test
* Having had a myocardial infarction
* Having had a cerebrovascular accident
* Having a rheumatological disease
* Known endocrine disease (Diabetes Mellitus, Hypo/hyperthyroidism)
* Cervical disc herniation defining radiculopathy
* Active trigger point palpated in the shoulder girdle muscles
* Having had any shoulder surgery
* Concomitant history of active systemic inflammatory disease, active infection and active malignancy
* Physical Therapy modalities have been applied in the last 6 months
* Having had an interventional procedure performed on the shoulder area within the last 6 months
* Using medications that may cause tendinopathy (Fluoroquinolines)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will be carried out cross-sectionally and in a single center, with patients diagnosed with Parkinson's disease who apply to the Physical Medicine and Rehabilitation Polyclinic of the University of Health Sciences Sultan 2.Abdülhamid Han Training and Research Hospital, and healthy volunteers who describe pain in any shoulder and who do not describe pain in any shoulder. The number of samples was calculated with G-power.Total of 160 patients and 320 shoulders were calculated.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
USG FINDINGS | ONE MONTH
  Measurements will be made by a Physical Medicine and Rehabilitation assistant physician experienced in musculoskeletal system ultrasonography, using the images obtained with the Sonosite M-Turbo device using the ImageJ program. During the measurements, the device will be positioned on the postero-lateral side of the patient while the patient and the practitioner are face to face. Five standard viewing windows will be used for the shoulder joint. These are: anterior transverse, anterior longitudinal, lateral longitudinal, lateral transverse, posterior transverse.

CONTACTS AND LOCATIONS:
Overall Officials: MEHMET AKİF GÜLER, Ass. Prof., Study Director — SULTAN ABDÜLHAMIDHAN TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided